CLINICAL TRIAL: NCT02805790
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Crossover Study to Evaluate Safety, Tolerability, and Efficacy of Subcutaneous Injections of MTP-131 in Subjects With Mitochondrial Myopathy Previously Treated in the SPIMM-201 Study
Brief Title: Safety, Tolerability, Efficacy of MTP-131 for Treatment of Mitochondrial Disease in Subjects From the MMPOWER Study
Acronym: MMPOWER-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPIMM-202
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Primary Mitochondrial Disease
Keywords: Primary Mitochondrial Disease; Mitochondrial Myopathy; Elamipretide; MTP-131; Bendavia™
MeSH Terms: conditions — Mitochondrial Myopathies | interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elamipretide, Then Placebo (Experimental): Participants first received 40 mg of elamipretide once daily subcutaneously for 4 weeks. After a washout period of 4 weeks, they then received placebo administered once daily subcutaneously for 4 weeks.
  Interventions: Drug: Elamipretide; Drug: Placebo
- Placebo, Then Elamipretide (Placebo Comparator): Participants first received placebo once daily subcutaneously for 4 weeks. After a washout period of 4 weeks, they then received 40 mg of elamipretide once daily subcutaneously for 4 weeks.
  Interventions: Drug: Elamipretide; Drug: Placebo

INTERVENTIONS:
Drug: Elamipretide — 4 weeks of treatment with 40 mg elamipretide administered once daily subcutaneously
  Other Names: Bendavia; MTP-131
Drug: Placebo — 4 weeks of treatment with placebo administered once daily subcutaneously

SUMMARY:
This randomized, double-blind, placebo-controlled, crossover study screened 32 subjects with primary mitochondrial myopathy (PMM) to evaluate the safety, tolerability, pharmacokinetics (PK), and efficacy of subcutaneous elamipretide in this patient population.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, crossover study screened 32 subjects with primary mitochondrial myopathy (PMM) who had completed participation in the SPIMM-201 study where they had received 5 days of intravenous (IV) elamipretide (0.01, 0.10, or 0.25 mg/kg/hour infused for 2 hours) or placebo (randomized 3:1). The primary objective was to evaluate the effect of single daily subcutaneous (SC) doses of elamipretide administered for 4 weeks on the 6-minute walking distance (6MWD).

Subjects were randomized (1:1) to one of two sequence groups: 4-weeks of treatment with 40 mg elamipretide administered once daily SC in Treatment Period 1 followed by 4-weeks of treatment with placebo administered once daily SC in Treatment Period 2 (separated by a 4-week washout period), or vice versa. Each sequence group went through 5 distinct periods: Screening, Treatment Period 1, Washout, Treatment Period 2, and Follow-Up. Safety, tolerability, pharmacokinetics (PK), and efficacy of subcutaneous elamipretide in this patient population were analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed participation in the SPIMM-201 study without a significant protocol deviation that would suggest the subject may not be able to complete all study requirements in the opinion of the Sponsor
* Subject must reside in North America for the duration of the study
* Subject has not received study drug in the SPIMM-201 study within 3 weeks prior to Screening
* Women of childbearing potential must agree to use 1 of the methods of birth control specified in the protocol from the date they sign the informed consent form (ICF) until two months after the last dose of study drug
* Subject has been on stable (unchanged and constant) medications (including over-the counter treatments, vitamins, or supplements) for at least 1 month prior to the Baseline Visit

Exclusion Criteria:

* Subject has any prior or current medical condition that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all study requirements (i.e. unstable angina or recent myocardial infarction)
* Subject has received any investigational compound and/or has participated in another interventional clinical study within 30 days prior to the Baseline Visit or is concurrently enrolled in any non-interventional research of any type judged to be scientifically or medically incompatible with the study as deemed by the Investigator in consultation with the Sponsor
* Subject experienced an adverse reaction to study drug in the SPIMM-201 study that contraindicates further treatment with elamipretide in the opinion of the Investigator and/or Sponsor
* Female subjects who are pregnant, planning to become pregnant, or lactating
* Subject has undergone an in-patient hospitalization within the 1 month prior to the Screening Visit or is likely to need in-patient hospitalization or a surgical procedure during the course of the study
* Subject has a creatinine clearance ≤30 mL/min as calculated by the Cockcroft Gault equation
* Subject has a corrected QT interval (QTc) elongation defined as a QTc >450 msec in male subjects and >480msec in female subjects. Note: At the initial electrocardiogram (ECG), if QTc exceeds these parameters, the ECG may be repeated 2 more times, and the average of the 3 QTc values used to determine the subjects eligibility
* Subject has uncontrolled hypertension in the judgment of the Investigator (e.g. elevated above >160 mmHg systolic or >100 mmHg diastolic despite appropriate treatment on two consecutive readings)
* Subject has a history of clinically significant hypersensitivity or allergy to any of the excipients contained in the study drug
* Subject has a history of active alcoholism or drug addiction during the year before the Screening Visit

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-08-22 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Carr, Study Director — Stealth BioTherapeutics
Locations (4):
- United States (4):
  - University of California, San Diego, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Akron Children's Hospital, Akron, Ohio
  - Children's Hospital of Pittsburg of UPMC, Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Gwaltney C, Stokes J, Aiudi A, Mazar I, Ollis S, Love E, Karaa A, Houts CR, Wirth RJ, Shields AL. Psychometric performance of the Primary Mitochondrial Myopathy Symptom Assessment (PMMSA) in a randomized, double-blind, placebo-controlled crossover study in subjects with mitochondrial disease. J Patient Rep Outcomes. 2022 Dec 23;6(1):129. doi: 10.1186/s41687-022-00534-y. PMID 36562873

RESULTS

PARTICIPANT FLOW:
Groups:
- Elamipretide, Then Placebo: Participants first received 40 mg of elamipretide once daily subcutaneously for 4 weeks. After a washout period of 4 weeks, they then received placebo administered once daily subcutaneously for 4 weeks.
  Elamipretide: 40 mg elamipretide administered once daily subcutaneously
Period: First Intervention (4 Weeks)
Arm/Group | Elamipretide, Then Placebo | Placebo, Then Elamipretide
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Washout (4 Weeks)
Arm/Group | Elamipretide, Then Placebo | Placebo, Then Elamipretide
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Elamipretide, Then Placebo | Placebo, Then Elamipretide
Started | 14 | 16
Completed | 14 | 15
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elamipretide, Then Placebo | Placebo, Then Elamipretide | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (16.67) | 48.6 (9.68) | 45.3 (13.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 15 | 25
  Male | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 13 | 16 | 29
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 22.8 (5.19) | 25.3 (5.46) | 24.1 (5.39)

OUTCOME MEASURES:

1. Primary Outcome: Distance Walked on the 6-minute Walk Test (6MWT) by Visit
Description: Distance in meters walked on the 6-minute walk test (6MWT) at end of treatment, where end of treatment means end of week 4 for Period 1 and end of week 12 for Period 2.
Time Frame: End of Week 4 and End of Week 12
Population: All participants for whom the distance walked on the 6MWT was measured.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Elamipretide: Participants who received 40mg Elamipretide administered once daily subcutaneously either the first or the last 4 weeks of the study.
- Placebo: Participants who received Placebo administered once daily subcutaneously either the first or the last 4 weeks of the study.
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 29 | 30
meters | 394.1 (134.16) | 378.2 (125.10)

2. Secondary Outcome: Wrist Accelerometer Counts by Day
Description: Wrist Accelerometer Counts by the last 7 days prior to the date of the end of treatment visit; End of treatment being end of Week 4 for Treatment Period 1 and end of Week 12 for Treatment Period 2. Subjects wore an activity monitor, or wrist accelerometer, on their wrist daily (from the Screening Visit to the End-of-Study/Early Discontinuation Visit). As a measure of physical activity and mobility, subjects wore an activity monitor, or wrist accelerometer, which measured mean vector magnitude of accelerations per daywith higher counts indicating a more active status. Raw acceleration data was converted into proprietary counts which was used to estimate physical activity. The data was transformed from 30 Hz data into 1 minute epoch data; this 1 minute epoch data were used for the analysis of as the vector magnitude of the wrist data.
Time Frame: Last 7 days prior to the date of end of treatment visit
Population: All participants for whom wrist accelerometer counts by day was measured.
Measure: Mean (Standard Deviation); unit: counts by day
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 30 | 29
counts by day | 1329.4 (505.28) | 1286.3 (507.83)

3. Secondary Outcome: Average Hip Accelerator Counts by Day
Description: Average Hip Accelerator Counts by last 7 days predose, and prior to end of treatment; End of treatment being Week 4 for Treatment Period 1 and Week 12 for Treatment Period 2. As a measure of physical activity and mobility, subjects wore an activity monitor, or hip accelerometer, on their hip (or belt line) daily during waking hours (minimum of at least 7 consecutive days immediately prior to study drug administration in each Treatment Period [Predose; at Visit 2 for Treatment Period 1 and at Visit 4 for Treatment Period 2]), and at the end of each Treatment Period [at Visit 3 for Treatment Period 1 and Visit 5 for Treatment Period 2]), which measured average acceleration per day, with higher counts indicating a more active status. Raw acceleration data was converted into proprietary counts which was used to estimate physical activity. The data was transformed from 30 Hz data into 1 minute epoch data; this 1 minute epoch data was used for the analysis of mean vertical axis (Y) cou
Time Frame: Last 7 days prior to the date of end of treatment visit
Population: All participants for whom hip accelerometer counts by day was measured.
Measure: Mean (Standard Deviation); unit: counts by day
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 30 | 30
counts by day
  Predose | 384.2 (130.70) | 380.6 (126.43)
  End of Treatment | 150.6 (162.13) | 148.1 (115.04)

4. Secondary Outcome: Neuro-QoL Fatigue Short Form Score: Total T-Scores (Question 1-8)
Description: Participants respond to the following statements of the Quality of Life in Neurological Disorders Fatigue Assessment (Neuro-QOL Fatigue Item Bank at end of treatment: I felt exhausted;I felt that I had no energy; I felt fatigued; I was too tired to do my household chores;I was too tired to leave the house;I was frustrated by being too tired to do the things I wanted to do; I felt tired; I had to limit my social activity because I was tired.Individual response options range from a score of 1 to 5, where 1=Never, 2=Rarely, 3=Sometimes, 4=Often, and 5=Always for end of treatment, where end of treatment period is end of week 4 for period 1, and end of week 12 for period 2. Raw scores are calculated as simple summed scores to an Item Response Theory Metric referred to as the T-score metric. Higher T-score means more fatigue, which means a worse outcome, with possible scores ranging from 29.5 to 74.1. Mean population T-score and standard deviation was reported.
Time Frame: End of Week 4 and End of Week 12
Population: All participants for whom Neuro-QoL Fatigue Short Form Score was measured.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 29 | 30
T-score | 50.9 (7.69) | 54.7 (10.35)

5. Secondary Outcome: Primary Mitochondrial Myopathy Symptom Assessment (PMMSA) Total Fatigue Score by Week
Description: Primary Mitochondrial Myopathy Symptom Assessment (PMMSA) Total Fatigue score at end of treatment (sum of Q1 to Q4; tiredness/muscle weakness) is scored as follows: 1=Not at all, 2=Mild, 3=Moderate, and 4=Severe. Total score range is 4-16; lower score means less fatigue and better outcome, higher score means more fatigue and worse outcome. Participants rate the following: Tiredness at rest, Tiredness during activities, Muscle weakness at rest, Muscle weakness during activities, at the end of each treatment period, where end of treatment period is the weekly average of the last 7 days of week 4 for period 1 and the last 7 days of week 12 for period 2.
Time Frame: Last 7 days of Week 4 and Last 7 days of Week 12
Population: All participants for whom PMMSA was measured at end of treatment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 30 | 30
score on a scale | 9.1 (2.35) | 10.7 (2.88)

6. Secondary Outcome: Triple Timed Up and Go (3TUG) Test by Visit
Description: Participant performed 3TUG test after the 6MWT, and after at least 15 minutes rest prior to study drug administration in each Treatment Period (End of Week 4 for Period 1 and End of Week 12 for Period 2.) Participant was directed to stand up from chair, walk at normal pace to the line on the floor 3 meters away,turn, walk back to the chair at normal pace, sit down again; activity was timed, in seconds. Activity is repeated 3 times consecutively without rest and an average time is calculated.
Time Frame: End of Week 4 and End of Week 12
Population: All participants for whom the 3TUG test was measured.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 29 | 30
seconds | 35.3 (16.66) | 35.2 (15.79)

7. Secondary Outcome: Patient Global Assessment [PGA] Score by Visit, Continuous
Description: Patient-reported current health status at end of treatment, where end of treatment means End of Week 4 for Period 1 and End of Week 12 for Period 2. PGA Scale is as follows: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Higher score means worse health status, means worse outcome.
Time Frame: End of Week 4 and End of Week 12
Population: All participants for whom the Patient Global Assessment was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 29 | 30
score on a scale | 3.4 (0.91) | 3.7 (1.01)

8. Secondary Outcome: Patient Global Assessment by Visit, Categorical
Description: Patient-reported current health status at end of treatment, where end of treatment means End of Week 4 for Period 1 and End of Week 12 for Period 2. PGA Scale is as follows: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Higher score means worse health status, means worse outcome. Excellent means excellent health, means better outcome; poor means poor health, means worse outcome.
Time Frame: End of Week 4 and End of Week 12
Population: All participants for whom the Patient Global Assessment was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 29 | 30
Participants
  Excellent | 1 | 1
  Very Good | 2 | 2
  Good | 12 | 8
  Fair | 11 | 12
  Poor | 3 | 7

9. Secondary Outcome: Physician Global Assessment (PhGA) By Visit, Continuous
Description: Physician Global Assessment (PhGA) Physician-reported overall health status at end of treatment, where end of treatment means End of Week 4 for Period 1 and End of Week 12 for Period 2.: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Higher scores equal worse outcome.
Time Frame: End of Week 4 and End of Week 12
Population: All participants for whom the Physician Global Assessment was measured.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 29 | 30
score on a scale | 3.1 (0.80) | 3.3 (0.84)

10. Secondary Outcome: Physician Global Assessment (PhGA) By Visit, Categorical
Description: Physician Global Assessment (PhGA) Physician-reported overall health status at end of treatment, where end of treatment means End of Week 4 for Period 1 and End of Week 12 for Period 2.: 1=Excellent, 2=Very good, 3=Good, 4=Fair, and 5=Poor. Higher scores equal worse outcome. Excellent means excellent health, means better outcome; poor means poor health, means worse outcome.
Time Frame: End of Week 4 and End of Week 12
Population: All participants for whom the Physician Global Assessment was measured.
Measure: Count of Participants; unit: Participants
Arm/Group | Elamipretide | Placebo
Number analyzed (Participants) | 29 | 30
Participants
  Excellent | 0 | 0
  Very Good | 6 | 5
  Good | 17 | 13
  Fair | 4 | 10
  Poor | 2 | 2

ADVERSE EVENTS:
Time Frame: Participants were followed for a total of 14 weeks; they had a Treatment Period for 4 weeks, then had a Washout Period of 4 weeks, then another Treatment Period of 4 weeks, then a Follow Up Period of 2 weeks.
Groups:
- Elamipretide: Participants received 40 mg of elamipretide once daily subcutaneously for 4 weeks, either in the first 4 weeks of treatment, or in the last 4 weeks of treatment.
- Placebo: Participants received placebo once daily subcutaneously for 4 weeks, either in the first 4 weeks of treatment or the last 4 weeks of treatment.
Arm/Group | Elamipretide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 30/30 | 15/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Elamipretide (N=30) | Placebo (N=30)
Injection site erythema (General disorders) | 17 | 1
Injection site pruritus (General disorders) | 14 | 0
Injection site pain (General disorders) | 6 | 1
Injection site urticaria (General disorders) | 6 | 0
Injection site bruising (General disorders) | 2 | 2
Injection site irritation (General disorders) | 3 | 1
Urinary Tract Infection (Infections and infestations) | 2 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 2 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Dizziness (Nervous system disorders) | 3 | 1
Dysarthria (Nervous system disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may not submit for publication or presentation the results of this study without first receiving written authorization from Stealth BioTherapeutics Inc. Stealth BioTherapeutics Inc., agrees that before it publishes any results of the study, it shall provide the Investigator with at least 30 days for review of the pre-publication manuscript prior to the submission of the manuscript to the publisher.

DOCUMENTS (2):
  • Study Protocol (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT02805790/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-21): https://cdn.clinicaltrials.gov/large-docs/90/NCT02805790/SAP_001.pdf